CLINICAL TRIAL: NCT03745430
Title: Phase Ib-II Study of Ramucirumab Combined With Standard Nab-paclitaxel and Gemcitabine as First-line Treatment in Patients With Advanced Pancreatic Adenocarcinoma
Brief Title: RAmucirumab Combined wIth Standard Nab-paclitaxel and Gemcitabine as First-line Chemotherapy in Patients With Advanced Pancreatic Adenocarcinoma
Acronym: RACING
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: Eli Lilly and Company (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE3/16; 2017-004792-30 (EudraCT Number)
Record Dates: First submitted 2018-11-07; First posted 2018-11-19 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ramucirumab+Nab-paclitaxel+Gemcitabine (Experimental): Nab-paclitaxel and Gemcitabine will be administered on days 1, 8 and 15 every 4 weeks for a maximum of 8 cycles.
  Interventions: Drug: Ramucirumab

INTERVENTIONS:
Drug: Ramucirumab — 8 mg/kg (days 1 and 15, q4w) until disease progression
  Other Names: Cyramza

SUMMARY:
RACING (RAmucirumab Combined wIth standard Nab-paclitaxel and Gemcitabine as first-line chemotherapy in patients with advanced pancreatic adenocarcinoma) trial is a Greek, investigator-initiated, single-arm, open-label phase Ib-II study. Patients with advanced cytologically or histologically proven pancreatic adenocarcinoma will be treated with a combination of Ramucirumab with Nab-paclitaxel and Gemcitabine (for a maximum of 8 cycles followed by Ramucirumab maintenance) until disease progression or excessive Adverse Events (AEs) or Investigator's decision or patient's refusal of further treatment or death, whichever comes first.

DETAILED DESCRIPTION:
Phase Ib: The first 12 patients will enter the phase Ib study in 2 cohorts of 6 patients each. In the first cohort, six patients will start Ramucirumab followed by Nab-paclitaxel and Gemcitabine every 4 weeks for 2 cycles at the specific initial dose level.When the dose is determined in the first cohort, then the second cohort will be enrolled to test the safety of this dose. The Phase II Recommended dose (RD) for the phase II part of the study will be determined when all 6+6 patients will complete a maximum of 2 cycles.

Phase II: In the phase II part of the trial, new patients will be recruited and start the study treatment according to the RD determined at the second cohort of the phase Ib part. Phase Ib patients will enter the phase II part by continuing the treatment beyond the second cycle at the RD level. All the patients will continue the treatment until disease progression or excessive AEs or completion of 8 cycles of Nab-paclitaxel/Gemcitabine/Ramucirumab. In patients with no progressive disease, ramucirumab monotherapy will be administered after the completion of 8 cycles of chemotherapy.

The primary endpoint will be Objective Response Rate (ORR) by RECIST criteria. Secondary endpoints will be Safety, Progression-free survival (PFS) and Overall Survival (OS). All the phase II endpoints will be assessed during BOTH the phase Ib and the phase II parts of the study. Patients enrolled at the phase Ib part will start being assessed for efficacy endpoints (response rate, PFS, OS) from the first date of registration to the study and will continue being assessed for efficacy also after passing to the phase II part of the study in a seamless way. After completion of patient enrollment in the phase Ib part, new patients will be enrolled directly to the phase II part. These patients will start being assessed for efficacy endpoints again from the first day of registration to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent
2. Histologically or cytologically proven pancreatic adenocarcinoma.
3. Metastatic or locally advanced unresectable disease confirmed clinically/radiologically by CT-scan or MRI (Magnetic Resonance Imaging)
4. No prior therapy for metastatic disease.
5. At least one measurable or evaluable lesion as assessed by CT-scan or MRI according to RECIST v1.1
6. Age 18 years,
7. ECOG Performance status (PS) 0-1
8. The patient has adequate hepatic function as defined by a total bilirubin 1.5 mg/dL (25.65 μmol/L), and aspartate transaminase (AST) and alanine transaminase (ALT) 2.5 times the upper limit of normal (ULN; or 5.0 times the ULN in the setting of liver metastases)
9. Female patients must commit to using reliable and appropriate methods of contraception during the trial until at least three months after the end of study treatment (when applicable). Male patients with a partner of childbearing potential must agree to use contraception in addition to having their partner use another reliable contraceptive method during the trial until at least 6 months after the end of study treatment.
10. Patients must have a low or intermediate risk of arterial or venous thrombotic events (Khorana risk score 0-2). Patients at a high VTE risk (Khorana RS3) are eligible if they receive LMWH prophylaxis (Appendix D).

Exclusion Criteria:

1. The patient has pancreatic cancer with histology other than adenocarcinoma
2. Prior therapy for metastatic disease. Adjuvant Gemcitabine is permitted if 6 or more months have elapsed from last cycle to date of relapse.
3. Exclusive presence of bone metastasis only
4. Concomitant unplanned antitumor therapy
5. Treatment with any other investigational medicinal product within 28 days prior to study entry
6. Other serious and uncontrolled non-malignant chronic disease
7. The patient has documented brain metastases, leptomeningeal disease, or uncontrolled spinal cord compression.
8. The patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal antiinflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325mg/day) is permitted.
9. The patient has experienced grade 3-4 gastrointestinal bleeding (unless due to resected tumor), treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, or diverticulitis within 3 months prior to first dose of protocol therapy.
10. Other concomitant or previous malignancy
11. The patient has symptomatic congestive heart failure (CHF; New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia
12. Bowel obstruction
13. The patient has a prior history of GI perforation/fistula (within 6 months of first dose of protocol therapy) or risk factors for perforation.
14. Palliative radiation therapy within 4 weeks prior to registration
15. The patient has a history of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy.
16. High risk for arterial or venous thrombotic complications as depicted by a Khorana Risk Score higher than 2 and inability to receive prophylaxis with low molecular weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Assessment of safety by identifying the Recommended Dose (RD) of the combination of Ramucirumab with Nabpaclitaxel and Gemcitabine. | From enrollment up to 90 days after the last administration of any investigational product
Phase II: Overall Response Rate is defined as the proportion of patients with confirmed Complete Response or confirmed Partial Response as best overall response to treatment, based on RECIST v. 1.1 guidelines in the considered analysis population. | Up to 33 months

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 33 months
Progression-free survival | Every 8 weeks until month 8 and then every 12 weeks, up to 33 months
Phase I:Toxicity profile of the combination during the first 2 cycles of therapy | From the first administration of study treatment and up to week 8 (during the first 2 cycles of the treatment, each cycle is 28 days)
Phase II: Number of participants with Serious and Non-Serious Adverse Events graded according to National Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 | From enrollment up to 33 months.
Investigation of SPARC gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of PTEN gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of MEK gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of AREG gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of EREG gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of VEGF-A gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of VEGF-B gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of PlGF gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of TSP1 gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of MMP2 gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of MMP9 gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months
Investigation of VEGFR1-3 gene mutation, m-RNA and protein expression | At baseline, in cycles 1 and 3 (each cycle is 28 days), at maintenance therapy and at the date of first documented progression up to 33 months

CONTACTS AND LOCATIONS:
Overall Officials: George Papaxoinis, MD, Principal Investigator — 2nd Medical Department, Agios Savvas Anticancer Hospital
Locations (13):
- Greece (13):
  - Agios Savvas Anticancer Hospital, Athens, Attica
  - Aretaieio Hospital, Athens, Attica
  - "Attikon" University Hospital, Chaïdári, Attica
  - Metropolitan General Hospital, Cholargós, Attica
  - Metropolitan Hospital, Neo Faliro, Attica
  - Ygeia Hospital, Psychikó, Attica
  - 3rd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens, Nea Kifisia
  - Agii Anargiri Cancer Hospital, Athens, Nea Kifisia
  - University Hospital of Patra, Rio, Patra
  - EUROMEDICA General Clinic of Thessaloniki, Thessaloniki, Thessaloniki
  - Haematology- Oncology Section, Dept of Clinical Therapeutics, General Hospital of Athens "Alexandra", Athens
  - Department of Medical Oncology, Ioannina University Hospital, Ioannina
  - General University Hospital of Larissa, Larissa